CLINICAL TRIAL: NCT05374239
Title: A Theory-driven Approach to Embed and Integrate a Post-stroke Upper Extremity Outcome Measure in Routine Clinical Practice
Brief Title: Embedding the Fugl-Meyer Assessment in Occupational Therapists' Routine Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Sengkang General Hospital (Other); Sengkang Community Hospital (Unknown); Outram Community Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: CIRB 2021/2559
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Implementation Science; Stroke
Keywords: implementation; outcome measures; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Hospital will be the unit of randomisation.
Who Masked: Participant
Masking Description: Due to the nature of intervention, blinding may not be possible. However, occupational therapists at all 4 hospitals will be blinded to the allocation sequence, with only the next hospital randomised for rollout being revealed at each intervention implementation time point. This will allow for blinding to the intervention partially possible. The investigators will also remind occupational therapists at all 4 hospitals not disclose details about the intervention to other healthcare professionals until the end of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hospital 1 (Other): First hospital in the allocation sequence to cross from control to intervention arm.
  Interventions: Other: Multi-component implementation intervention
- Hospital 2 (Other): Second hospital in the allocation sequence to cross from control to intervention arm.
  Interventions: Other: Multi-component implementation intervention
- Hospital 3 (Other): Third hospital in the allocation sequence to cross from control to intervention arm.
  Interventions: Other: Multi-component implementation intervention
- Hospital 4 (Other): Fourth hospital in the allocation sequence to cross from control to intervention arm.
  Interventions: Other: Multi-component implementation intervention

INTERVENTIONS:
Other: Multi-component implementation intervention — The multiple-component implementation intervention will comprise of 3 key components: (1) education, (2) operational process, and (3) audit and feedback

SUMMARY:
Background: Using outcome measures is emphasized in foundational training and clinical practice guidelines, but less than 50% of rehabilitation professionals consistently use outcome measures in practice. No studies have evaluated the barriers to routine outcome measurement in Singapore's healthcare settings nor identified effective implementation strategies to sustain the use of outcome measures in practice.

Aims: To evaluate the effectiveness of a tailored multi-component implementation intervention effectiveness in improving the consistency of use of the Fugl-Meyer Assessment of Upper Extremity (FMA) among occupational therapists practicing in 4 hospitals in Singapore.

Method: The project will use the Normalisation Process Theory as a framework and data collection sites will include Singapore General Hospital, Sengkang General Hospital, Outram Community Hospital, and Sengkang Community Hospital. The investigators will use a stepped-wedge randomised trial design. The study will begin with an initial period in which no hospitals are exposed to the intervention. Subsequently, at regular intervals, one hospital will cross from the control to the intervention. The investigators will continue this process until the intervention is introduced to all hospitals. The intervention will be fully implemented by the end of the trial, with all 4 hospitals receiving the multi-component intervention.

Project Significance: This trial is part of a larger project that uses a theory-driven approach to systematically explore the embedding and integration of outcome measures in routine clinical care for rehabilitation professionals in Singapore (beyond initial implementation stages). Study findings will contribute to the scientific knowledge base of implementing outcome measures in clinical practice, improve patient care, and support future implementation projects on outcome measurement in different populations and healthcare settings.

DETAILED DESCRIPTION:
Study Hypothesis:

The null hypothesis is there is no change in the average rate of adherence to the administration to the FMA 6 months post-intervention. The alternate hypothesis is there is a significant improvement in the average rate of adherence to the administration of the FMA 6 months post-intervention.

Study Design:

The investigators will use a stepped-wedge randomized trial to evaluate the effectiveness of the implementation strategy (i.e. intervention), which involves a sequential crossover of hospitals from the control to the intervention arm (Figure 3). The study will begin with an initial period in which no hospitals are exposed to the intervention. Subsequently, at regular intervals (2 month duration), one hospital will cross from the control to the intervention. The investigators will continue this process until the intervention is introduced to all hospitals. The intervention will be fully implemented by the end of the trial, with all 4 hospitals receiving the intervention. The trial will include the 4 hospitals based on convenience sampling.

Intervention:

This trial will be conducted as part of a larger research project that uses a theory-driven approach to systematically explore the embedding and integration of outcome measures in routine clinical care for rehabilitation professionals in Singapore. The multi-component implementation strategy (i.e. intervention) will be developed in earlier phases of the larger project.

Outcomes:

The primary endpoint will be the average rate of adherence to the administration of the FMA 6 months post-intervention.

Randomisation:

Hospital will be the unit of randomisation. The investigators will employ simple randomisation using concealed envelopes.

Blinding:

Due to the nature of intervention, blinding may not be possible. However, occupational therapists at all 4 hospitals will be blinded to the allocation sequence, with only the next hospital randomised for rollout being revealed at each intervention implementation time point. This will allow for blinding to the intervention partially possible. The investigators will also remind occupational therapists at all 4 hospitals not disclose details about the intervention to other healthcare professionals until the end of the trial.

ELIGIBILITY:
A total of 4 acute and hospitals will be part of the study. These hospitals were identified through convenience sampling based on the following criteria:

Inclusion Criteria:

* Affiliated to SingHealth
* Currently using FMA in clinical practice by occupational therapists

Exclusion Criteria:

* Use of FMA in clinical practice by occupational therapists funded by existing research grants
* Not using FMA in clinical practice by occupational therapists

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Adherence rate | 6 months post-intervention
  Average rate of adherence to the administration of the FMA by occupational therapists

OTHER OUTCOMES:
Acceptability of Intervention Measure (AIM) | 6 months post-intervention
  Brief 4-item pragmatic measure of implementation outcome. Each item is rated on a 5-point ordinal scale.
Intervention Appropriateness Measure (IAM) | 6 months post-intervention
  Brief 4-item pragmatic measure of implementation outcome. Each item is rated on a 5-point ordinal scale.
Feasibility of Intervention Measure (FIM) | 6 months post-intervention
  Brief 4-item pragmatic measure of implementation outcome. Each item is rated on a 5-point ordinal scale.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Choo, PhD, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No